CLINICAL TRIAL: NCT06053749
Title: INFORM - Interferon-Beta Exposure in the 2nd and 3rd Trimester of Pregnancy - a Register-Based Drug Utilisation Study in Finland and Sweden
Brief Title: An Observational Study to Learn About the Interferon-beta Exposure of Pregnant Women During the Second and Third Trimester in Finland and Sweden
Acronym: INFORM
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Biogen Netherlands B.V (Unknown); Novartis Europharm Limited (Unknown); Merck Europe B.V. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21334; EUPAS38736 (Other: ENCEPP)
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis (MS)
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a; Interferon beta-1b; peginterferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pregnancies exposed to IFNB only: With dispensed IFNB, no other MS disease modifying drugs (MSDMDs) during the pre-pregnancy period or during pregnancy
  Interventions: Drug: Avonex (IFNβ-1-a, Biogen Netherlands B.V); Drug: Rebif (IFNβ-1-a, Merck Europe B.V.); Drug: Extavia (IFNβ-1-b, Novartis Europharm Limited); Drug: Betaseron (IFN-β-1-b, BAY86-5046, Bayer AG); Drug: Plegridy (Peg IFNβ-1-a, Biogen Netherlands B.V)
- Pregnancies unexposed to IFNB nor other MSDMDs: No dispensed IFNB nor any other MSDMDs during the pre-pregnancy period nor any time during pregnancy
- Pregnancies exposed to IFNB (regardless of other MSDMDs): With dispensed IFNB, regardless of other MS disease modifying drugs (MSDMDs) during the pre-pregnancy period or during pregnancy
  Interventions: Drug: Avonex (IFNβ-1-a, Biogen Netherlands B.V); Drug: Rebif (IFNβ-1-a, Merck Europe B.V.); Drug: Extavia (IFNβ-1-b, Novartis Europharm Limited); Drug: Betaseron (IFN-β-1-b, BAY86-5046, Bayer AG); Drug: Plegridy (Peg IFNβ-1-a, Biogen Netherlands B.V); Drug: MS disease modifying drugs (MSDMDs)
- Pregnancies unexposed to IFNB (regardless of other MSDMDs): No dispensed IFNB during the pre-pregnancy period nor any time during pregnancy, regardless of other MSDMDs
  Outcomes:
  Interventions: Drug: MS disease modifying drugs (MSDMDs)

INTERVENTIONS:
Drug: Avonex (IFNβ-1-a, Biogen Netherlands B.V) — Information on drug use in hospitals and outpatient clinics are not recorded in the drug registers used in the study and, thus, information on exposure to these medications is not available.
  Groups: Pregnancies exposed to IFNB (regardless of other MSDMDs); Pregnancies exposed to IFNB only
Drug: Rebif (IFNβ-1-a, Merck Europe B.V.) — Information on drug use in hospitals and outpatient clinics are not recorded in the drug registers used in the study and, thus, information on exposure to these medications is not available.
  Groups: Pregnancies exposed to IFNB (regardless of other MSDMDs); Pregnancies exposed to IFNB only
Drug: Extavia (IFNβ-1-b, Novartis Europharm Limited) — Information on drug use in hospitals and outpatient clinics are not recorded in the drug registers used in the study and, thus, information on exposure to these medications is not available.
  Groups: Pregnancies exposed to IFNB (regardless of other MSDMDs); Pregnancies exposed to IFNB only
Drug: Betaseron (IFN-β-1-b, BAY86-5046, Bayer AG) — Information on drug use in hospitals and outpatient clinics are not recorded in the drug registers used in the study and, thus, information on exposure to these medications is not available.
  Groups: Pregnancies exposed to IFNB (regardless of other MSDMDs); Pregnancies exposed to IFNB only
Drug: Plegridy (Peg IFNβ-1-a, Biogen Netherlands B.V) — Information on drug use in hospitals and outpatient clinics are not recorded in the drug registers used in the study and, thus, information on exposure to these medications is not available.
  Groups: Pregnancies exposed to IFNB (regardless of other MSDMDs); Pregnancies exposed to IFNB only
Drug: MS disease modifying drugs (MSDMDs) — Information on drug use in hospitals and outpatient clinics are not recorded in the drug registers used in the study and, thus, information on exposure to these medications is not available.
  Groups: Pregnancies exposed to IFNB (regardless of other MSDMDs); Pregnancies unexposed to IFNB (regardless of other MSDMDs)

SUMMARY:
Observational data have suggested no increased risk of adverse pregnancy outcomes associated with exposure to interferon-beta (IFNB) before or during pregnancy. After the emergence of these data, the European Medicines Agency approved a label change for IFNB in September 2019, stating that use of IFNB during pregnancy may be considered, if clinically needed. However, limited data on pregnancies exposed in the 2nd and 3rd trimesters were observed.

INFORM is a secondary use of data drug utilisation study (DUS) to determine late pregnancy exposure (i.e. during the 2nd and 3rd trimester) to IFNB in Finland and Sweden, which will inform whether the number of exposed pregnancies is adequate to conduct a cohort study on adverse pregnancy outcomes, with a focus on late pregnancy exposure.

The number of pregnancies will be initially reported three years after the revised label implementation (September 2019) and will include data on pregnancies from 1996 in Finland and from 2005 in Sweden up through 31 December 2022. If the number of pregnancies is deemed adequate for conducting the cohort study on adverse pregnancy outcomes, this DUS will be finalised with the drug utilisation data accrued up through 31 December 2022. If the number of pregnancies until 31 December 2022 is deemed inadequate, this study may be continued and the primary and secondary objectives may be examined five years after the revised label implementation, including pregnancies until 31 December 2024.

ELIGIBILITY:
Inclusion Criteria:

* Women with a diagnosis of MS disease, regardless of MS clinical type, recorded at least once during the full study period.
* Women with at least one recorded pregnancy after the MS diagnosis (including pregnancies ending in live birth, stillbirth, spontaneous abortion, ectopic pregnancy, or elective termination)

Exclusion Criteria:

- None.

Ages: 12 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Aggregate secondary data will be collected from the following national registers in Finland and Sweden.
  FINLAND: Medical Birth Register (MBR-Fin), Care Register for Health Care, National Reimbursement Register/National Prescription Register, Register of Induced Abortions.
  SWEDEN: Medical Birth Register (MBR-Swe), National Patient Register (NPR), Swedish Prescribed Drug Register (SPDR).
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The number of pregnancies of women with MS, not allowing exposure to other MS Disease Modifying Drugs (MSDMDs) | Data recorded between 01 January 1996 - 31 December 2022 in Finland, and 01 July 2005 - 31 December 2022 in Sweden.
  Analysis groups: Pregnancies exposed to IFNB only group and Pregnancies unexposed to IFNB nor other MSDMDs group
The level of precision for the risk of pre-defined adverse pregnancy outcomes in late pregnancy that can be obtained with the available number of exposed and unexposed pregnancies | Data recorded between 01 January 1996 - 31 December 2022 in Finland, and 01 July 2005 - 31 December 2022 in Sweden.
  Pre-defined adverse pregnancy outcomes:
  * Anomalies: Major congenital anomalies (MCA); All anomalies, including minor and major
  * Fatal outcomes: Spontaneous abortions, Elective terminations, Stillbirth and Neonatal mortality
  * Growth outcomes: Small for gestation age and Low birth weight
  * Other outcomes: Preterm birth
  Late pregnancy, i.e. the 2nd and 3rd trimester.
The annual number of pregnancies of women with MS in the exposure groups | Data recorded between 2015-2019 and 2020-2022.
  Analysis in Pregnancies exposed to IFNB only group.

SECONDARY OUTCOMES:
The number of pregnancies of women with MS in Finland and Sweden in exposure groups allowing exposure to other MSDMDs | Data recorded between 01 January 1996 - 31 December 2022 in Finland, and 01 July 2005 - 31 December 2022 in Sweden.
  Analysis groups: Pregnancies exposed to IFNB (regardless of other MSDMDs) group and Pregnancies unexposed to IFNB (regardless of other MSDMDs) group
The annual number of women with MS in childbearing age, and with dispensed IFNB | Data recorded between 2015 to 2022 in Finland and Sweden

CONTACTS AND LOCATIONS:
Locations (2):
- Many locations, Multiple Locations, Finland
- Many locations, Multiple Locations, Sweden

IPD SHARING:
Plan to Share IPD: No
No data will be shared

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/